CLINICAL TRIAL: NCT04343183
Title: Hyperbaric Oxygen Therapy (HBOT) as a Treatment for COVID-19 (COVID-19) Infection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive IRB approval
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001051
Record Dates: First submitted 2020-04-07; First posted 2020-04-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: This study will utilize a single-center sequential two-parallel-group (HBOT/Standard care) randomized controlled design with 2 looks to allow for early stop due to clear benefit/harm.
Who Masked: Outcomes Assessor
Masking Description: The biostatistician and radiologist will not know which group received HBOT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HBOT treatment group (Active Comparator): Patients will receive hyperbaric oxygen therapy
  Interventions: Device: Hyperbaric Oxygen Therapy
- Standard of Care group (No Intervention): Patients will not receive hyperbaric oxygen therapy and will receive the current standardized treatment protocol

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy delivered at a specific uniformed pressure and duration.
  Arms: HBOT treatment group

SUMMARY:
Patients who meet inclusion criteria will be randomized into treatment vs control group. Treatment groups will undergo Hyperbaric Oxygen Therapy (HBOT) and compared to the control group.

DETAILED DESCRIPTION:
After enrollment, patients will be randomized into treatment vs control group. Both populations will receive the same inpatient medical treatment. All patients in the treatment group will undergo hyperbaric oxygen therapy under the same treatment protocol. After completion of the treatment protocol, specific study endpoints will be compared between the treatment and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients >18 years old
* Positive PCR COVID-19 testing
* CT evidence of interstitial opacity
* Oxygen saturation <90% on room air
* pO2 = 55-70.

Exclusion Criteria:

* Increased oxygen requirements
* Hemodynamic instability (MAP<65)
* Bradycardia (HR<50)
* History of seizure disorder
* Pneumothorax
* GFR<30
* Hemodialysis
* Refractory anxiety/claustrophobia
* Current pregnancy
* Uncorrectable hypoglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Decrease incidence of intubation by 30% or greater | one month
  Compare rates of intubation between treatment and control groups

SECONDARY OUTCOMES:
Decrease renal injury | one month
  Measure Glomerular Filtration Rate (GFR) and compare between treatment and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery S Kuo, MD, Study Chair — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Participants will be given a unique unidentifiable study ID number and all data will be recorded accorded to unidentifiable number to protect the patients personal health information.